CLINICAL TRIAL: NCT04620018
Title: Comparison of Three Antibiotic Protocols in Prevention of Infection in Dental Implant Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shiraz University of Medical Sciences (Other)
Collaborators: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Principal Investigator, RTabrizi, Shiraz university of medical sciences, Shiraz University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1399
Record Dates: First submitted 2020-11-02; First posted 2020-11-06 (Actual); Last update posted 2020-11-20 (Actual); Status verified 2020-11

CONDITIONS: Dental Implant Failed
Keywords: dental implant; osseointegration; infection
MeSH Terms: conditions — Infections | interventions — Amoxicillin; halofantrine

STUDY DESIGN:
Intervention Model Description: subjects were aligned randomly into three groups.In group 1, subjects received prophylactic antibiotic orally (Amoxicillin 2mg ,1 hour before surgery) and post-surgical antibiotic (Amoxicillin 500 mg , q8h for five days), subjects received only prophylactic antibiotic (Amoxicillin 2mg ,1 hour before surgery) in group 2 ,and in group 3, subjects received post-surgical antibiotic (Amoxicillin 500 mg , q8h for five days) .
Who Masked: Participant
Masking Description: An independent investigator who was blind to participants (groups) evaluated all subjects
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Pre and post op Antibiotic (Active Comparator): subjects received prophylactic antibiotic orally (Amoxicillin 2mg ,1 hour before surgery) and post-surgical antibiotic (Amoxicillin 500 mg , q8h for five days)
  Interventions: Drug: Amoxicillin
- Pre-op antibiotic (Active Comparator): subjects received only prophylactic antibiotic (Amoxicillin 2mg ,1 hour before surgery)
  Interventions: Drug: Amoxicillin
- Post-op antibiotic (Active Comparator): subjects received post-surgical antibiotic (Amoxicillin 500 mg , q8h for five days)
  Interventions: Drug: Amoxicillin

INTERVENTIONS:
Drug: Amoxicillin — Subjects received Amoxicillin before surgery, before and after surgery ,and only after surgery.
  Other Names: GLAXOSMITHKLINE

SUMMARY:
Subjects who underwent a dental implant surgery were studied.Subjects randomly were aligned into three groups:In group 1, subjects received prophylactic antibiotic orally (Amoxicillin 2mg ,1 hour before surgery) and post-surgical antibiotic (Amoxicillin 500 mg , q8h for five days), subjects received only prophylactic antibiotic (Amoxicillin 2mg ,1 hour before surgery) in group 2 ,and in group 3, subjects received post-surgical antibiotic (Amoxicillin 500 mg , q8h for five days). The sign and symptom of infection were studied and the incidence of infection in each group was determined.

DETAILED DESCRIPTION:
Subjects eligible for study inclusion had an edentulous area in the mandible or maxilla and underwent a dental implant surgery. Subjects were excluded from study enrollment if they had systemic diseases which affect bone metabolism, history of allergy to amoxicillin, refused study enrollment or failed to return for follow-up.

Subjects were randomly divided into three groups : In group 1, subjects received prophylactic antibiotic orally (Amoxicillin 2mg ,1 hour before surgery) and post-surgical antibiotic (Amoxicillin 500 mg , q8h for five days), subjects received only prophylactic antibiotic (Amoxicillin 2mg ,1 hour before surgery) in group 2 ,and in group 3, subjects received post-surgical antibiotic (Amoxicillin 500 mg , q8h for five days) . An independent researcher made random allocation cards using computer-generated random. Then, allocated cases were placed in a sealed envelope. All subjects used 0.2% chlorhexidine mouthwash in the treatment period. All implants were placed with a two-stage protocol.

All subjects were followed up for 3 months to assess any infection signs and symptoms. Infection was diagnosed based on clinical findings such as pain, redness of the area, and discharge around the fixture.An independent dentist who was blind the study groups, evaluated all subjects.

ELIGIBILITY:
Inclusion Criteria:

* Have an edentulous area in the mandible or maxilla
* underwent a dental implant surgery

Exclusion Criteria:

* systemic diseases which affect bone metabolism
* history of allergy to amoxicillin
* refused study enrollment
* failed to return for follow-up.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 450 (Actual)
Dates: Start 2016-09-30 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
Infection incidence | 3 months
  pain, redness of the area, and discharge around the fixture.

CONTACTS AND LOCATIONS:
Overall Officials: Reza Tabrizi, DDS, Study Director — Shiraz University of Medical Sciences

IPD SHARING:
Plan to Share IPD: Yes
We can present the data of participant without individual identification.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: 12.1.2020
Access Criteria: Researchers who are eligible to access shahid beheshti university of medical sciences website
URL: http://sbmu.ac.ir